CLINICAL TRIAL: NCT00382915
Title: Nicotine Intake in Smokers With Schizophrenia
Brief Title: Measuring Smoking Behavior in People With Schizophrenia and Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: R01MH076672 (NIH); R01MH076672 (NIH); DAHBR 96-BHB
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Smoking; Topography; Nicotine
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for DNA extraction
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Smokers with schizophrenia
  Interventions: Device: CReSSmicro handheld topography device
- 2: Smokers with bipolar disorder
  Interventions: Device: CReSSmicro handheld topography device
- 3: Smokers without any mental illness
  Interventions: Device: CReSSmicro handheld topography device

INTERVENTIONS:
Device: CReSSmicro handheld topography device — The CReSS micro device represents the state-of-the-art technology for measurements of ambulatory puff topography taken in the smoker's natural environment. Although all topography measurements are limited, at least to some degree, by the artificial act of smoking while using a device, or smoking through a mouthpiece, this small, lightweight and portable device is easy to use outside of the laboratory setting to capture more naturalistic smoking behavior and allows for less intrusion from the research team and research environment.

SUMMARY:
This study will evaluate the differences in smoking behavior, nicotine intake, and nicotine boost among people with schizophrenia, bipolar disorder, or no mental illness.

DETAILED DESCRIPTION:
People with schizophrenia, a disabling mental disorder, smoke at rates three times higher than those of the general population. They also tend to develop serious medical problems due to this heavy smoking. Little is known, however, about the relationship between schizophrenia and smoking. Smoking topography, the study of cigarette-puffing behavior, may help to uncover important information about the smoking habits of people with schizophrenia, and how they differ from smokers who do not have a mental illness. To develop more effective treatment approaches for schizophrenic smokers, a better understanding of nicotine addiction in this population is needed. This study will use hand-held smoking topography devices and blood tests to measure smoking behavior and nicotine levels in people with schizophrenia. This information will be compared to similar measurements in people with no mental illness and in people with bipolar disorder, another disorder associated with high rates of heavy smoking.

Participation in this open-label, observational study will last approximately 1 to 2 weeks, and will consist of two to three study visits. The first visit will last about 2 hours, and will include screening procedures, completion of baseline questionnaires, and a practice session of smoking topography. Subjects will return on a second day (Day 2) for the remainder of the study procedures to assess their smoking puffing behavior and nicotine intake from usual cigarette smoking, which will occur within 1 week of the Day 1 assessments. On the afternoon prior to Day 2 subjects will have a brief appointment to review instructions for using the topography device. They will take the topography with them and be instructed to use it as they smoke ad-lib that evening at home. This will serve as a second practice session for getting used to the topography device. They will also be instructed to use the device for all cigarettes smoked upon awakening the next day at 6am (Day 2), including the first cigarette of the day. They will go to the study site for the first of three blood tests at 9:30 A.M, after which they will be allowed to leave the study site to continue with their daily activities. They will use the smoking topography device throughout the day, until 3 P.M. At this time, study staff will go to each participant's location to collect the device. Participants will have two additional blood tests over the course of the study to measure nicotine levels.

ELIGIBILITY:
Inclusion Criteria:

For smokers with schizophrenia or bipolar disorder:

* Meets DSM-IV diagnostic criteria for schizophrenia or bipolar I disorder
* Smokes 10 or more cigarettes every day
* Has been stable on current psychiatric medications for at least 1 month prior to study entry

For control smokers without mental illness:

* Smokes 10 or more cigarettes every day

Exclusion Criteria:

For smokers with schizophrenia or bipolar disorder:

* Current or past suicidal ideation, behavior, or suicide attempt within 30 days prior to study entry
* Psychiatric hospitalization within 30 days prior to study entry
* Inability to read English or inability to sufficiently understand study documents written in English
* Pregnant, breastfeeding, or plans to become pregnant within 1 month of study entry
* Current use of any non-cigarette forms of tobacco (e.g., cigars, pipes, smokeless tobacco, or ultralight cigarettes)
* Current substance abuse problem, as defined by DAST or AUDIT criteria
* Significant cognitive impairment that may interfere with study participation, as defined by a Folstein Mini-Mental Status exam score of less than 22

For control smokers without mental illness:

* Any DSM-defined mental disorder within 1 year prior to study entry
* Inability to read English or inability to sufficiently understand study documents written in English
* Concomitant use of nicotine replacement therapy (e.g., gum, patch, inhaler, nasal spray, or lozenge), clonidine, bupropion, or nortriptyline
* Pregnant, breastfeeding, or plans to become pregnant within 1 month of study entry
* Current use of any non-cigarette forms of tobacco (e.g., cigars, pipes, smokeless tobacco, or ultralight cigarettes)
* Diagnosis or treatment for an episode of any mental disorder (e.g., depression or anxiety) within 1 year prior to study entry
* Lifetime diagnosis of bipolar disorder or schizophrenia
* Lifetime history of any psychotic symptoms
* Lifetime use of antipsychotic medication for any reason
* Use of any antidepressants, mood stabilizers, or anti-anxiety medications for any reason within 6 months prior to study entry
* Current substance abuse problem, as defined by DAST or AUDIT criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be 100 smokers with schizophrenia, 100 smokers with bipolar disorder and 100 smokers without mental illness. This will include smokers within the New Jersey metropolitan area, who receive treatment at the UMDNJ-University Behavioral Health Care System (UBHC) or at another outpatient behavioral health care agency. A community sample of healthy volunteer smokers without mental illness will be recruited through advertisements to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2006-10; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Smoking behavior and nicotine levels in those diagnosed with schizophrenia, those diagnosed with bipolar disorder and, those without a current mental illness | Measured at Hour 24

SECONDARY OUTCOMES:
Difference in blood levels of cotinine in smokers with schizophrenia compared to controls | Measured at Hour 24

CONTACTS AND LOCATIONS:
Overall Officials: Jill M. Williams, MD, Principal Investigator — Rutgers, The State University of New Jersey; Kunal K. Gandhi, MBBS, MPH, Study Director — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ-Robert Wood Johnson Medical School, Department of Psychiatry, Division of Addictions, New Brunswick, New Jersey, United States

REFERENCES:
- [Result] Williams JM, Gandhi KK, Lu SE, Kumar S, Steinberg ML, Cottler B, Benowitz NL. Shorter interpuff interval is associated with higher nicotine intake in smokers with schizophrenia. Drug Alcohol Depend. 2011 Nov 1;118(2-3):313-9. doi: 10.1016/j.drugalcdep.2011.04.009. Epub 2011 May 18. PMID 21596491
- [Result] Williams JM, Gandhi KK, Benowitz NL. Carbamazepine but not valproate induces CYP2A6 activity in smokers with mental illness. Cancer Epidemiol Biomarkers Prev. 2010 Oct;19(10):2582-9. doi: 10.1158/1055-9965.EPI-10-0384. Epub 2010 Aug 18. PMID 20719908
- [Result] Williams JM, Gandhi KK, Lu SE, Kumar S, Shen J, Foulds J, Kipen H, Benowitz NL. Higher nicotine levels in schizophrenia compared with controls after smoking a single cigarette. Nicotine Tob Res. 2010 Aug;12(8):855-9. doi: 10.1093/ntr/ntq102. Epub 2010 Jun 28. PMID 20584771